CLINICAL TRIAL: NCT01348958
Title: Evaluation of Orthopedic Knee Measurement Using Lunar iDXA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 105-2011-GES-0001-000
Record Dates: First submitted 2011-05-02; First posted 2011-05-06 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Hemi Knee Arthroplasty; Patello-femoral Osteoarthritis
Keywords: Patello femoral; osteoarthritis; arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post-operative knee replacement (Experimental): Subjects that have had a hemi knee replacement of one knee at least 8 weeks ago had the post-operative knee scanned using the orthopedic hip application and the Lunar orthopedic knee application.
  Interventions: Device: iDXA knee software

INTERVENTIONS:
Device: iDXA knee software — Following surgery, subjects who have undergone knee arthroplasty will have the knee that has undergone arthroplasty (post-operative) scanned at least 8 weeks after surgery.
  During one visit, each subject will have the post-operative knee scanned 1 time using Lunar orthopedic application, and 3 times with the subject repositioned between scans using the Lunar orthopedic knee application (total of 4 scans). Lunar iDXA measurement procedures will be done
  Other Names: DXA; iDxa

SUMMARY:
This study is to compare scans of the knee performed using new software designed specifically to look at the knee joint with those performed using approved software designed for scans of the hip.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>30 years) males and females.
2. Have had a hemi knee replacement of one knee at least 8 weeks ago.
3. Patello-femoral osteoarthritis is not a contraindication if person does not have symptoms from the patello-femoral joint.
4. Able to provide informed consent.
5. In good general health.

Exclusion Criteria:

1. Neuromuscular or vascular disease in the affected leg.
2. Found to be unsuitable for hemi knee arthroplasty (KA) before or at surgery.
3. Preoperative extensions defect greater than 15 degrees.
4. Preoperative maximal flexion of less than 100 degrees.
5. Symptomatic patello-femoral osteoarthritis.
6. Insufficiency of anterior cruciate ligament (ACL)
7. Fracture sequalae (Intraarticular fracture and all tibial condyle fractures).
8. Previous osteotomy.
9. Previous extensive knee surgery.
10. Metabolic bone disease including osteoporosis with a T score of <-2.5.
11. Rheumatoid arthritis.
12. Postmenopausal women on systemic hormone replacement therapy (HRT).
13. Long-term treatment with oral corticosteroids and/or bisphosphonates.
14. Inability to consent (such as Alzheimer's Disease).
15. Misuse of drugs or alcohol.
16. Serious psychiatric disease.
17. Disseminated malignant disease and treatment with radiotherapy or chemotherapy.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of Lunar orthopedic knee software. | 5 months from starting study.
  This study will compare the bone density and bone mass measurements acquired with Lunar orthopedic knee software and for the same scans acquired with Lunar orthopedic software. A determination of precision of bone measurements acquired and analyzed with Lunar orthopedic knee software.

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Gilchrist, M.D., Principal Investigator — CGM Reseach Trust - Princess Margaret Hospital
Locations (1):
- CGM Research Trust - Princess Margaret Hospital, Cashmere, Christchurch, New Zealand